CLINICAL TRIAL: NCT05647473
Title: Efficacy, Safety and Response Predictors of Adjuvant Astragalus for Cognition in Alzheimer Disease With Orthostatic Hypotension: an add-on, Assessor-blind, Pragmatic Randomized Controlled Trial
Brief Title: Efficacy, Safety and Response Predictors of Adjuvant Astragalus for Cognition in Orthostatic Hypotension
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AM-AD
Record Dates: First submitted 2022-12-04; First posted 2022-12-12 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Orthostatic Hypotension; Alzheimer Disease
MeSH Terms: conditions — Hypotension, Orthostatic; Alzheimer Disease

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- add-on low dose Astragalus (Experimental)
  Interventions: Behavioral: Routine treatment; Drug: add-on low dose Astragalus
- Routine treatment (Experimental)
  Interventions: Behavioral: Routine treatment
- add-on high dose Astragalus (Experimental)
  Interventions: Behavioral: Routine treatment; Drug: add-on high dose Astragalus

INTERVENTIONS:
Behavioral: Routine treatment — Participants will be educated on ways to avoid induced hypotensive states, such as avoiding prolonged standing, standing after exercise, being nervous, eating several carbohydrate-rich foods, drinking alcohol, and being in a warm environment (such as a sauna). Participants will be encouraged in a comfortable home environment, such as a sit-down bath. If there are no contraindications, they are advised to increase their salt intake to approximately 10 grams per day and adjust their fluid intake to 2-3 liters per day. They will also be encouraged to perform lower-body strength training and moderate, non-strenuous activities. Seriously ill patients will be proposed to raise the head of their bed during sleep, wear tight clothing, eat small meals, and reduce alcohol intake.Concomitant treatment with cholinesterase inhibitors, memantine, or both was allowed.
Drug: add-on low dose Astragalus — Participants received an additional 10g of astragalus per day.
  Arms: add-on low dose Astragalus
Drug: add-on high dose Astragalus — Participants received an additional 20g of astragalus per day.
  Arms: add-on high dose Astragalus

SUMMARY:
Background: This pragmatic clinical trial aims to determine the efficacy and safety of add-on Astragalus for cognition and non- cognition in patients with of mild to moderate Alzheimer's disease complicated with orthostatic hypotension in orthostatic hypotension, elucidate the underlying mechanisms, identify related response predictors, and explore effective drug components.

Methods: This is an add-on, assessor-blinded, parallel, pragmatic, randomized controlled trial. At least 66 adults with mild to moderate Alzheimer's disease (AD) and OH aged >30 years will be recruited. Participants will be randomized in a 1:1:1 ratio to receive 24 weeks of routine care or add-on low dose Astragalus or high dose Astragalus group. The primary efficacy outcome will be measured by the Alzheimer's Disease Assessment Scale-Cognitive Subscale, Chinese version. Secondary efficacy outcome assessment will include neuropsychological tests, blood pressure, plasma biomarkers, multimodal electroencephalograms, and neuroimaging. Safety outcome measures will include physical examinations, vital signs, electrocardiography, laboratory tests (such as hematologic and blood chemical tests), and adverse event records.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria will be as follows:

1. Male or female aged ≥50 years and ≤85 years
2. A decrease in systolic blood pressure of 20 mm Hg or a decrease in diastolic blood pressure of 10 mm Hg within 3 minutes after standing.
3. Memory loss for at least 6 months, with a progressive worsening trend
4. Patients with mild or moderate disease degree, that is, the total score of MMSE: 14 points < total score of MMSE <24 points, 0.5≤CDR≤2 points, and the total score of HAMD (24-item version) ≤20 points
5. Brain magnetic resonance imaging shows the degree of hippocampal atrophy is greater than or equal to grade 1
6. The modified Hachinski Ischemia Scale (m-HIS) score was < 4 points
7. The criteria described by the diagnostic and statistical manual of mental disorder-V for the diagnosis of dementia comply with the National Institute on Aging - Alzheimer's Association "Very likely AD" (National Institute of Aging-Alzheimer's Association, 2011).
8. There are no obvious positive signs in nervous system examination;
9. The subjects have the ability of reading, writing and communication, have a stable caregiver, accompany to attend the visit.
10. The basic treatment of AD before enrollment remained unchanged, and if long-term users needed to use it steadily for more than 4 weeks before randomization,the dose was kept as stable as possible during the study. Such drugs include: cholinesterase inhibitors and diamantine.

Exclusion Criteria:

The exclusion criteria will be as follows:

1. MRI showed significant focal lesions, including one of the following: a. There were more than 2 infarcts with a diameter greater than 2cm; b. Infarcts in key areas such as the thalamus, hippocampus, entorhinal cortex, parorhinal cortex, angular gyrus, cortex, and other subcortical gray matter nuclei; c. White matter lesion Fazekas Scale ≥3
2. Patients who have taken other Chinese medicine preparations in the past three months
3. Allergy or contraindication of astragalus
4. There are other neurological diseases that can cause brain dysfunction or cognitive impairment; Mental and neurological retardation is present; Presence of malignant tumor
5. The modified Hachinski Ischemia Scale (m-HIS) score was ≥ 4 points.
6. Patients who refuse or have MRI or EEG contraindications (pacemakers, coronary and peripheral arterial stents, Metal implants, claustrophobia, or severe visual or hearing impairment), refusing to draw blood
7. Pregnant or lactating patients;
8. Patients who have participated in other clinical studies within the past 3 months

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-02-20 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
The primary efficacy outcome measure will be the absolute change in the Alzheimer's Disease Assessment Scale-Cognitive Subscale, Chinese version score between baseline and week 48. | Participants will be followed up for 48 weeks after baseline.
  The Alzheimer's Disease Assessment Scale-Cognitive Subscale, Chinese version scale scores range from 0 to 75, with higher scores indicating better.

SECONDARY OUTCOMES:
The absolute scores change in the Rey-Osterrieth Complex Figure Test [ROCF] recall score between baseline and week 48. | Participants will be followed up for 48 weeks after baseline.
  The ROCF scale scores range from 0 to 36, with higher scores indicating better.
The absolute scores change in the ROCF-copy score between baseline and week 48. | Participants will be followed up for 48 weeks after baseline.
  The ROCF copy scale scores range from 0 to 36, with higher scores indicating better.
The absolute scores change in the Clock-Drawing Test score between baseline and week 48. | Participants will be followed up for 48 weeks after baseline.
  The Clock-Drawing Test scale scores range from 0 to 5, with higher scores indicating better.
The absolute scores change in the Trail Making Test-A score between baseline and week 48. | Participants will be followed up for 48 weeks after baseline.
  The Trail Making Test-A scores range from 0 to 25, with higher scores indicating better.
The absolute scores change in the Digit Span Forward score between baseline and week 48. | Participants will be followed up for 48 weeks after baseline.
  TheDigit Span Forward score scores range from 0 to 10, with higher scores indicating better.
The absolute scores change in the Trail Making Test-B score between baseline and week 48. | Participants will be followed up for 48 weeks after baseline.
  The Trail Making Test-B scores range from 0 to 25, with higher scores indicating better.
The absolute scores change in the Digit Span Backward score between baseline and week 48. | Participants will be followed up for 48 weeks after baseline.
  TheDigit Span Forward score scores range from 0 to 9, with higher scores indicating better.
The absolute scores change in the Verbal Fluency Test score between baseline and week 48. | Participants will be followed up for 48 weeks after baseline.
  The Verbal Fluency Test score scores range from 0 to 14, with higher scores indicating better.
The absolute scores change in the Hamilton Anxiety Scale score between baseline and week 48. | Participants will be followed up for 48 weeks after baseline.
  The Hamilton Anxiety Scale score scores range from 0 to 56, with higher scores indicating worse.
The absolute scores change in the Hamilton Depression Scale score between baseline and week 48. | Participants will be followed up for 48 weeks after baseline.
  The Hamilton Anxiety Scale score scores range from 0 to 96, with higher scores indicating worse.
The absolute change in the blood pressure between baseline and week 48. | Participants will be followed up for 48 weeks after baseline.
  To observe the changes of orthostatic blood pressure in patients
The absolute change in the level of plasma β-amyloid40 (ng/ml) between baseline and week 48. | Participants will be followed up for 48 weeks after baseline.
  Amyloid is one of the main biomarkers of dementia
The absolute change in the level of plasma β-amyloid42 (ng/ml) between baseline and week 48. | Participants will be followed up for 48 weeks after baseline.
  Amyloid is one of the main biomarkers of dementia
The absolute change in the level of plasma glial fibrillary acidic protein (ng/ml) between baseline and week 48. | Participants will be followed up for 48 weeks after baseline.
  Glial fibrillary acidic protein is one of the main biomarkers of dementia
The absolute change in the level of plasma neurofilament light chain (ng/ml) between baseline and week 48. | Participants will be followed up for 48 weeks after baseline.
  Neurofilament light chain is one of the main biomarkers of dementia
The absolute change in the level of plasma hyper-phosphorylated tau-181 (ng/ml) between baseline and week 48. | Participants will be followed up for 48 weeks after baseline.
  Neurofilament light chain is one of the main biomarkers of dementia
The absolute change in the P300 between baseline and week 48. | Participants will be followed up for 48 weeks after baseline.
  P300 is the main indicator of EEG, and its normal value range is between 320 and 420.
The absolute change in the VP300 between baseline and week 48. | Participants will be followed up for 48 weeks after baseline.
  VP300 is the main indicator of EEG, and its normal value range is between 320 and 420.
The absolute change in the MMN between baseline and week 48. | Participants will be followed up for 48 weeks after baseline.
  MMN is the main indicator of EEG, and its normal value range is between 100 and 210.
The absolute change in the neurite density index between baseline and week 48. | Participants will be followed up for 48 weeks after baseline.
  Neurite density index is the main indicator of neurite-oriented diffusion and density imaging (NODDI) .
The absolute change in the orientation dispersion index between baseline and week 48. | Participants will be followed up for 48 weeks after baseline.
  Orientation dispersion index is the main indicator of neurite-oriented diffusion and density imaging (NODDI) .
The absolute change in the isotropic volume fraction between baseline and week 48. | Participants will be followed up for 48 weeks after baseline.
  Isotropic volume fraction is the main indicator of neurite-oriented diffusion and density imaging (NODDI) .
The absolute change in theheart rate variability between baseline and week 48. | Participants will be followed up for 48 weeks after baseline.
  The KARDi2/4-B autonomic nervous function mapping ECG system (Nanjing Left and Right Brain Biomedical Company, NeuroMed, China) will record and analyze millivolt-level signals of ECG oscillations, complete the frequency domain and time domain index detection of heart rate variability in 3 min, and generate an autonomic nervous function status step map.
The absolute change in the Montreal Cognitive Assessment(MOCA) score between baseline and week 48. | Participants will be followed up for48 weeks after baseline.
  The Alzheimer's Disease Assessment Scale-Cognitive Subscale, Chinese version scale scores range from 0 to 30, with higher scores indicating better.

OTHER OUTCOMES:
Whether the participants' vital signs were normal. | Participants will be followed up for 48 weeks after baseline.
  Safety outcome
Whether the participants' Electrocardiograms were normal. | Participants will be followed up for 48 weeks after baseline.
  Safety outcome
Whether the participants' Liver function were normal. | Participants will be followed up for 48 weeks after baseline.
  Safety outcome
Whether the participants' kidney function were normal. | Participants will be followed up for 48 weeks after baseline.
  Safety outcome
Severity of adverse events | Participants will be followed up for 48 weeks after baseline.
  Safety outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cheng Y, Lin L, Huang P, Zhang J, Pan X. Efficacy, safety, and response predictors of Astragalus in patients with mild to moderate Alzheimer's disease: A study protocol of an assessor-blind, statistician-blind open-label randomized controlled trial. Contemp Clin Trials Commun. 2024 Jul 28;41:101339. doi: 10.1016/j.conctc.2024.101339. eCollection 2024 Oct. PMID 39176240